CLINICAL TRIAL: NCT01786590
Title: Endobronchial Ultrasound-guided Transbronchial Needle Aspiration for Lymph Node Staging in Patients With Non-small Cell Lung Cancer Pursuing Stereotactic Body Radiotherapy (SBRT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-5294-CE
Record Dates: First submitted 2013-02-04; First posted 2013-02-08 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EBUS-TBNA (Experimental)
  Interventions: Procedure: EBUS-TBNA

INTERVENTIONS:
Procedure: EBUS-TBNA — Currently EBUS-TBNA is performed in patients with CT and/or PET positive lymph nodes in the mediastinum or hilum. In this study, all patients being considered for SBRT will undergo EBUS-TBNA for the lymph node staging prior to SBRT.

SUMMARY:
It is reported that more than 90,000 patients died of lung cancer and more than 20% of them were older than 80 years in North America. Therefore a less invasive but effective treatment is required for patients with lung cancer of advanced age, diminished pulmonary functions, and chronic diseases. Stereotactic body radiation therapy (SBRT) is an effective and well-tolerated treatment for early stage lung cancer in medically inoperable patients. On the other hand, accurate mediastinal and hilar lymph node staging is one of the most important factors that determine the outcome and indications for SBRT. Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) is a novel, minimally invasive modality that enables the assessment of mediastinal and hilar lymph nodes with a high sensitivity. Accurate lymph node staging by EBUS-TBNA will allow opportunities for high-risk patients with lung cancer to undergo minimally invasive treatment.

DETAILED DESCRIPTION:
Patients with radiologically early stage lung cancer who are candidates for SBRT will be enrolled in this study. Prior to enrollment, patients are required to be evaluated by an experienced thoracic surgeon, radiation oncologist or medical oncologist to determine operability. Patients will udergo computed tomography (CT) and positron emission tomography (PET) prior to EBUS- TBNA. EBUS-TBNA will be performed at the Interventional Thoracic Surgery Suite (ITSS) located at Toronto General Hospital by a Thoracic Surgeon. The procedure will be performed under local anesthesia with conscious sedation. Mediastinal as well as hilar lymph nodes will be assessed by EBUS-TBNA. The result of pathological diagnosis using EBUS-TBNA will be compared with the result of radiological staging (CT and PET-CT). Patients who are negative for mediastinal lymph node metastasis by EBUS-TBNA will undergo SBRT. In addition, the treatment outcome will be evaluated based on the clinical chart review.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Patients with confirmed lung cancer who require EBUS-TBNA as part of their staging investigations of the mediastinum and hilum prior to SBRT
3. Performance status score (WHO/ECOG) of 0-2.
4. Cytological or histological proof of non-small cell cancer
5. Stage T1-2 disease, with no evidence of distant metastasis
6. Patients are screened by both computed tomography (CT) and positron emission tomography (PET)
7. Medically inoperable for surgical resection
8. Patients who refused surgery

Exclusion Criteria:

1. Patients who are deemed on clinical grounds not to be medically fit for a bronchoscopy
2. Active systemic, pulmonary, or pericardial infection
3. Patients who are pregnant or lactating
4. Patients with plans to receive conventional radiotherapy, chemotherapy, biological therapy, vaccine therapy, or surgery as treatment (except at disease progression).
5. Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-02; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To test whether or not there is a difference in accuracy between CT/PET and the minimally invasive technique of EBUS-TBNA for mediastinal staging in patients with non-small cell lung cancer prior to stereotactic body radiotherapy (SBRT). | 3 years
  Primary objective: To test whether or not there is a difference in accuracy between CT/PET and the minimally invasive technique of EBUS-TBNA for mediastinal staging in patients with non-small cell lung cancer prior to stereotactic body radiotherapy (SBRT).
  In comparing EBUS-TBNA vs. CT/PET the primary outcome measures will be:
  1) Sensitivity, 2) Specificity, 3) Positive predictive value, 4) Negative predictive value, 5) Accuracy in detecting malignancy

SECONDARY OUTCOMES:
The treatment outcome (nodal recurrence rate) will be evaluated based on clinical chart review. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Yasufuku, MD, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada